CLINICAL TRIAL: NCT01346189
Title: A Randomized Trial of Behavioral Economic Interventions to Reduce CVD Risk
Brief Title: A Trial of Behavioral Economic Interventions to Reduce Cardiovascular Disease (CVD) Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Geisinger Clinic (Other); Brigham and Women's Hospital (Other); Harvard School of Public Health (HSPH) (Other); Carnegie Mellon University (Other); Harvard Vanguard Medical Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 812701; RC4AG039114 (NIH)
Record Dates: First submitted 2011-04-26; First posted 2011-05-02 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-10

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Physician Incentives (Active Comparator): (with adherence feedback)
  Quarterly payments to physician combined based on patient achieving an LDL reduction of at least 10 mg/dl relative to baseline LDL or the last quarter's target LDL with daily patient statin adherence information made available.
  Interventions: Behavioral: Behavioral Economic Intervention
- Patient Incentives (Active Comparator): (with adherence feedback)
  Quarterly payments to patient based on patient achieving an LDL reduction of at least 10 mg/dl relative to baseline LDL or the last quarter's target LDL.
  Interventions: Behavioral: Behavioral Economic Intervention
- Physician and Patient Combined Incentives (Active Comparator): (with adherence feedback)
  Quarterly payments shared evenly by physician and patient based on patient achieving an LDL reduction of at least 10 mg/dl relative to baseline LDL or the last quarter's target LDL. Physicians will receive daily information about patients' statin adherence.
  Interventions: Behavioral: Behavioral Economic Intervention
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Behavioral Economic Intervention — Various combinations of financial incentives to patients and providers.
  Arms: Patient Incentives; Physician Incentives; Physician and Patient Combined Incentives

SUMMARY:
Using a 4-arm, cluster-randomized controlled trial, the investigators will test the effectiveness of different behavioral economic interventions in increasing statin use and reducing LDL cholesterol among patients with poor cholesterol control who are at very high risk for CVD. The investigators will test these approaches among primary care physicians and their patients at very high risk of CVD at Geisinger Health System and University of Pennsylvania outpatient clinics.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in the United States. Despite strong evidence that reducing low-density lipoproteins (LDL) with statins successfully lowers CVD risk, physicians under-prescribe statins, physicians fail to intensify treatment when indicated, and more than 50% of patients stop taking statins within one year of first prescription, though such therapy typically should be life-long. In this study, we will test the effectiveness of different behavioral economic interventions in increasing statin use and reducing LDL cholesterol among patients with poor cholesterol control who are at very high risk for CVD. The application of conceptual approaches from behavioral economics offers considerable promise in advancing health and health care. Pay for performance initiatives represent one such potential application, but one in which incorporating the underlying psychology of decision makers has not generally been done, and experimental tests have not been conducted. We will test these approaches among primary care physicians and their patients at very high risk of CVD at Geisinger Health System and University of Pennsylvania outpatient clinics. Using a 4-arm, cluster-randomized controlled trial, we aim to answer these questions: [1] How does the provision of provider incentives compare to the provision of patient incentives, to a combination of patient and provider incentives, or to no incentives at all? [2] Are results sustained after incentives and other interventions are withdrawn? [3] How do these approaches compare in implementation, acceptability, cost, and cost-effectiveness?

ELIGIBILITY:
Inclusion Criteria:

* Physicians: All primary care providers who have at least 5 patients who meet eligibility criteria will be eligible.
* Patients: 10-year CVD risk of between 10-20% who do not have an LDL below 140 mg/dl or 10-year CVD risk of at least 20% (including those with preexisting CHD) who do not have an LDL below 120 mg/dl will be the primary inclusion criteria. We have chosen to include all patients meeting these inclusion criteria regardless of their reported adherence to statins, as there clearly is room for improvement in the LDL through a combination of physician and patient actions.

Exclusion Criteria:

* Patients will be excluded if they have a known allergy or history of side effects to statins, will not or cannot give consent, or have a markedly shortened life expectancy (diagnosis of metastatic cancer, end-stage renal disease on dialysis, or dementia).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1503 (Actual)
Dates: Start 2011-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Volpp, MD, PhD, Principal Investigator — University of Pennsylvania; David Asch, MD, MBA, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Harvard Vanguard Medical Associates, Boston, Massachusetts
  - Geisinger Health System, Danville, Pennsylvania
  - Unversity of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Rosenthal MB, Troxel AB, Volpp KG, Stewart WF, Sequist TD, Jones JB, Hirsch AG, Hoffer K, Zhu J, Wang W, Hodlofski A, Finnerty D, Huang JJ, Asch DA. Moderating Effects of Patient Characteristics on the Impact of Financial Incentives. Med Care Res Rev. 2019 Feb;76(1):56-72. doi: 10.1177/1077558717707313. Epub 2017 May 8. PMID 29148344
- [Derived] Asch DA, Troxel AB, Stewart WF, Sequist TD, Jones JB, Hirsch AG, Hoffer K, Zhu J, Wang W, Hodlofski A, Frasch AB, Weiner MG, Finnerty DD, Rosenthal MB, Gangemi K, Volpp KG. Effect of Financial Incentives to Physicians, Patients, or Both on Lipid Levels: A Randomized Clinical Trial. JAMA. 2015 Nov 10;314(18):1926-35. doi: 10.1001/jama.2015.14850. PMID 26547464

RESULTS

PARTICIPANT FLOW:
Groups:
- Physician Incentives: (with adherence feedback)
  Quarterly payments to physician combined based on patient achieving an LDL reduction of at least 10 mg/dl relative to baseline LDL or the last quarter's target LDL with daily patient statin adherence information made available.
  Behavioral Economic Intervention: Various combinations of financial incentives to patients and providers.
- Patient Incentives: (with adherence feedback)
  Quarterly payments to patient based on patient achieving an LDL reduction of at least 10 mg/dl relative to baseline LDL or the last quarter's target LDL.
  Behavioral Economic Intervention: Various combinations of financial incentives to patients and providers.
- Physician and Patient Combined Incentives: (with adherence feedback)
  Quarterly payments shared evenly by physician and patient based on patient achieving an LDL reduction of at least 10 mg/dl relative to baseline LDL or the last quarter's target LDL. Physicians will receive daily information about patients' statin adherence.
  Behavioral Economic Intervention: Various combinations of financial incentives to patients and providers.
- Usual Care/Control: No Intervention
Period: Overall Study
Arm/Group | Physician Incentives | Patient Incentives | Physician and Patient Combined Incentives | Usual Care/Control
Started | 433 | 358 | 346 | 366
Completed | 417 (433 patients (64 primary care physicians) included in analysis) | 341 (358 Patients (58 primary care physicians) included in analysis) | 332 (346 patients (58 primary care physicians) included in analysis) | 355 (366 patients (58 primary care physicians) included in analysis)
Not Completed | 16 | 17 | 14 | 11
Not completed — Withdrawal by Subject | 7 | 5 | 3 | 5
Not completed — Physician Decision | 4 | 0 | 0 | 0
Not completed — Moved | 3 | 0 | 4 | 0
Not completed — Other | 2 | 4 | 7 | 3
Not completed — Death | 0 | 3 | 0 | 0
Not completed — Non-health system primary care physician | 0 | 5 | 0 | 0
Not completed — Travel | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: No Intervention
- Total: Total of all reporting groups
Arm/Group | Physician Incentives | Patient Incentives | Physician and Patient Combined Incentives | Usual Care | Total
Number analyzed (Participants) | 433 | 358 | 346 | 366 | 1503
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.68 (8.67) | 62.41 (8.63) | 62.03 (8.64) | 61.70 (8.89) | 61.99 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179 | 164 | 135 | 161 | 639
  Male | 254 | 194 | 211 | 205 | 864
Race/Ethnicity [Count of Participants; unit: Participants]
  White, non-Hispanic | 360 | 265 | 285 | 289 | 1199
  African American, non-Hispanic | 57 | 72 | 42 | 61 | 232
  Other non-Hispanic | 8 | 10 | 6 | 7 | 31
  Hispanic | 6 | 10 | 7 | 7 | 30
  Missing | 2 | 1 | 6 | 2 | 11
Annual Household Income, No., $ [Count of Participants; unit: Participants]
  <50,000 | 193 | 145 | 134 | 163 | 635
  50,000 to 100,000 | 144 | 129 | 126 | 124 | 523
  >100,000 | 85 | 76 | 68 | 68 | 297
Education [Count of Participants; unit: Participants]
  <College | 148 | 107 | 102 | 129 | 486
  Some college | 118 | 102 | 108 | 105 | 433
  College and postcollege graduate | 165 | 148 | 133 | 131 | 577
Marital Status [Count of Participants; unit: Participants]
  Single | 64 | 59 | 43 | 59 | 225
  Married | 286 | 236 | 239 | 231 | 992
  Other | 81 | 62 | 60 | 75 | 278
Framingham Risk Score (FRS) [Mean (Standard Deviation); unit: %] — The Framingham Risk Score is a gender-specific algorithm used to estimate the 10-year cardiovascular risk of an individual. Individuals with low risk have 10% or less CHD risk at 10 years, with intermediate risk 10-20%, and with high risk 20% or more.
  % | 20.1 (9.0) | 19.7 (8.6) | 19.1 (8.7) | 20.1 (8.7) | 19.8 (8.7)
Pre-existing coronary artery disease (CAD) [Count of Participants; unit: Participants] | 143 | 110 | 115 | 148 | 516
Taking cholesterol-reducing medications at baseline [Count of Participants; unit: Participants] | 166 | 180 | 200 | 166 | 712

OUTCOME MEASURES:

1. Primary Outcome: Change in LDL From Baseline to 12 Months
Description: Change in LDL-C levels (mg/dL)
Time Frame: 12 months
Population: Subjects were lost to follow-up, or withdrawn for other reasons. Thus the number analyzed at the 12 month time point does not equal the number analyzed during baseline.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Physician Incentives | Patient Incentives | Physician and Patient Combined Incentives | Usual Care
Number analyzed (Participants) | 433 | 358 | 346 | 366
mg/dL
  Mean Reduction | 27.9 [24.9 to 31.0] | 25.1 [21.6 to 28.5] | 33.6 [30.1 to 37.1] | 25.1 [21.7 to 28.5]
  Baseline | 159.9 [157.4 to 162.5] | 160.6 [157.6 to 163.0] | 160.1 [157.3 to 163.3] | 161.5 [159.0 to 164.7]
  12 Months: number analyzed (Participants) | 396 | 329 | 317 | 331
  12 Months | 132 [127.8 to 135.3] | 135.5 [130.8 to 138.9] | 126.4 [123.1 to 130.1] | 136.4 [132.5 to 140.7]

2. Secondary Outcome: Change in LDL From Baseline to 15 Months
Description: Change in LDL-C levels (mg/dL) from baseline to 15 months
Time Frame: 15 months
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Physician Incentives | Patient Incentives | Physician and Patient Combined Incentives | Usual Care
Number analyzed (Participants) | 433 | 358 | 346 | 366
mg/dL | 29.1 [25.3 to 32.9] | 23.9 [19.8 to 27.9] | 32.8 [28.7 to 36.8] | 25.8 [21.5 to 30.2]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the subjects' participation in the study; 15 month time period.
Description: Defining Adverse Events:
  In this study, ALT greater than or equal to three times the upper limit of normal was considered an adverse event.
  Defining Serious Adverse Events:
  A definition for an SAE was assigned as ALT greater than or equal to 400 U/L, or hospitalizations or deaths caused by Myalgia or Rhabdomyolysis or liver toxicity.
Arm/Group | Physician Incentives | Patient Incentives | Physician and Patient Combined Incentives | Usual Care/Control
All-Cause Mortality (participants affected / at risk) | 2/433 | 3/358 | 0/346 | 1/366
Serious Adverse Events (participants affected / at risk) | 0/433 | 0/358 | 1/346 | 0/366
Other Adverse Events (participants affected / at risk) | 0/433 | 0/358 | 0/346 | 1/366
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physician Incentives (N=433) | Patient Incentives (N=358) | Physician and Patient Combined Incentives (N=346) | Usual Care/Control (N=366)
Pancreatic mass (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Follow up CT scan revealed a large pancreatic obstructing mass compressing the common bile duct. With this clinical picture, this is the most likely cause for the transaminase elevation, and not statin related, as verified by subject's PCP
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physician Incentives (N=433) | Patient Incentives (N=358) | Physician and Patient Combined Incentives (N=346) | Usual Care/Control (N=366)
Elevated Alanine Aminotransferase (ALT) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Elevated ALT lab result. ALT was determined by subject's PCP to not be study related; but rather due to methotrexate medication, which was stopped.

LIMITATIONS AND CAVEATS:
Patients in the control group received electronic pill bottles and may have been more adherent than is typical; Mean of about 6 patients per physician enrolled, limiting total size of potential reward; Adherence info came from pill bottle opening

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes